CLINICAL TRIAL: NCT06587425
Title: A Phase II Study Evaluating the Efficacy and Safety of LM-302 in Combination With Candonilimab and Capecitabine for First-Line Treatment in Patients With Unresectable Advanced, Recurrent, or Metastatic CLDN18.2-Positive Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: The Efficacy and Safety of LM-302 in Combination With Candonilimab and Capecitabine for First-Line Treatment in Patients With Unresectable Advanced, Recurrent, or Metastatic CLDN18.2-Positive Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Tianshu Liu, Professor, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LM-302-IIT-203
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gastric or Gastroesophageal Junction Adenocarcinoma
Keywords: CLDN18.2; ADC drug; cadonilimab; Immune Checkpoint Inhibitor; Targeted therapy; Immunotherapy; Chemotherapy

STUDY DESIGN:
Intervention Model Description: The study is divided into a safety lead-in phase and an expansion phase. The safety lead-in phase will evaluate the dose-limiting toxicity (DLT) of the LM-302 combined with cadonilimab and capecitabine regimen in patients with unresectable, recurrent, or metastatic CLDN18.2-positive gastric or gastroesophageal junction adenocarcinoma. Based on the safety data obtained from the lead-in phase, the expansion phase will determine the drug dosage and assess the efficacy and safety of the LM-302 combined with cadonilimab and capecitabine regimen in the same patient population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LM-302+Cadonilimab+Capecitabine (Experimental): LM-302: 1.8mg/kg ivgtt d1, q2w; Canonilimab: 6mg/kg ivgtt d1, q2w; Capecitabine: 1000mg/m^2 po bid d1-10, q2w.
  Interventions: Drug: LM-302+Candonilimab+Capecitabine

INTERVENTIONS:
Drug: LM-302+Candonilimab+Capecitabine — LM-302: 1.8mg/kg ivgtt d1, q2w; Canonilimab: 6mg/kg ivgtt d1, q2w; Capecitabine: 1000mg/m^2 po bid d1-10, q2w.
  Other Names: ADC-Claudin18.2+AK104+Capecitabine

SUMMARY:
A Phase II Study Evaluating the Efficacy and Safety of LM-302 in Combination with Candonilimab and Capecitabine for First-Line Treatment in Patients with Unresectable Advanced, Recurrent, or Metastatic CLDN18.2-Positive Gastric or Gastroesophageal Junction Adenocarcinoma

DETAILED DESCRIPTION:
The antibody-drug conjugate (ADC) targeting CLDN18.2 exerts its anti-tumor effects through multiple mechanisms, including direct cytotoxicity to CLDN18.2-positive tumor cells via the delivery of a potent small-molecule toxin, a bystander effect that induces cytotoxicity in adjacent CLDN18.2-negative tumor cells, and the activation of the immune system through antibody-dependent cellular cytotoxicity (ADCC). The combination of this ADC with immune checkpoint inhibitors holds potential for synergistic anti-tumor activity. LM-302, an ADC specifically targeting CLDN18.2 and comprising a monoclonal antibody conjugated to MMAE, has demonstrated favorable efficacy and safety profiles in both preclinical and clinical studies for CLDN18.2-expressing gastrointestinal malignancies, including gastric and gastroesophageal junction adenocarcinomas. The combination of LM-302 with immune checkpoint inhibitors may offer enhanced clinical benefits for patients with advanced gastric cancer.

This clinical study aims to evaluate the efficacy and safety of LM-302 (ADC targeting Claudin18.2) in combination with cadonilimab (a bispecific antibody targeting PD-1 and CTLA-4) and capecitabine as a first-line treatment in patients with unresectable, recurrent, or metastatic CLDN18.2-positive gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* The subjects fully understand the purpose, nature, methods, and potential adverse reactions of the trial, voluntarily participate as participants, and sign an informed consent form (ICF) before any procedures begin
* The subject must have locally advanced or metastatic gastric cancer or gastroesophageal junction cancer that cannot be surgically removed, and the histopathological examination confirms it to be simple adenocarcinoma
* Permissible Previous Treatment: Participants with gastric cancer or gastroesophageal junction cancer who have previously received adjuvant or neoadjuvant treatment and have experienced clinical disease progression at least 6 months after the last administration are eligible for inclusion. (Note: The treatment-related toxicity of oxaliplatin in previous adjuvant or neoadjuvant treatments must be restored to the National Cancer Institute [NCI] General Terminology Standard for Adverse Events [CTCAE] v5.0 Level 1 before enrollment)
* CLDN18.2 positivity: Provide sufficient tissue markers for Claudin18.2 immunohistochemistry testing. Claudin18.2 immunohistochemistry expression ≥ 10% is confirmed as positive, and<10% is recorded as negative
* According to RECIST v1.1 standard, there should be at least one measurable lesion
* ECOG physical state ≤ 1
* Expected lifespan>3 months
* Adequate renal function: creatinine (Cr) ≤ 1.5 x upper limit of normal (ULN) and glomerular filtration rate (GFR) ≥ 60mL/min/1.73 m2;
* Sufficient liver function: Total bilirubin ≤ 1.5 × ULN, AST and ALT ≤ 2.5 × ULN (if there is liver metastasis, AST and ALT ≤ 5 × ULN, total bilirubin ≤ 2.5 × ULN);
* Adequate bone marrow reserve: Platelet count (PLT) ≥ 100 × 109/L, absolute neutrophil count (ANC) ≥ 1.5 × 109/L, hemoglobin ≥ 9 g/dL (no adjuvant therapy such as EPO, G-CSF, or GM-CSF has been received within 14 days, and no blood transfusion including red blood cells and platelets has been received at least 7 days before the first administration); Prothrombin time/activated partial thromboplastin time (PT/PTT)<1.5 x ULN;
* Male or female aged ≥ 18 years old.

Exclusion Criteria:

* Known HER2 positive gastric cancer/adenocarcinoma of the gastroesophageal junction. HER2 positivity refers to HER2 amplification that requires confirmation from ISH if the HER2 immunohistochemistry test result is 3+and the immunohistochemistry test result is 2+
* Has undergone major surgery or radiation therapy within 4 weeks prior to enrollment;
* Active, known or suspected autoimmune diseases
* Congestive heart failure or symptomatic coronary artery disease within 3 months prior to enrollment
* A cerebrovascular accident occurred within the past 6 months
* Clinically significant bleeding, bleeding events, or thromboembolic diseases occur within 6 months
* History of intestinal perforation
* Have a history of (non infectious) pneumonia requiring steroid treatment or currently suffer from pneumonia
* Known history of human immunodeficiency virus (HIV) infection. Subjects with active hepatitis B or active hepatitis C. (Unless receiving antiviral therapy for at least 14 days prior to the first study drug administration and passing hepatitis B virus (HBV) DNA titer testing (not exceeding 500 IU/mL or 2500 copies [cps]/mL) and hepatitis C virus (HCV) RNA testing (not exceeding the lower limit of the assay), eligible for inclusion in the trial and willing to continue receiving effective antiviral therapy during the study period);
* Severe impairment of lung function or history of interstitial lung disease
* Diagnosed with concurrent malignant tumors within the past 2 years (except for fully treated non melanoma skin cancer, superficial bladder transitional cell carcinoma, and cervical carcinoma in situ [CIS]) or any currently active malignant tumor
* Previous or current evidence suggests that there may be confusion with the research results, interference with the participant's participation in the entire study process, any conditions, treatments, or laboratory abnormalities, or the researcher believes that participating in this study is not in the best interest of the participant
* Pregnancy test positive within 7 days before the first administration, or women of childbearing age who are in lactation period
* Individuals with known mental illnesses or disorders that may affect trial compliance
* Subjects who take systemic corticosteroids (>10 mg daily prednisone equivalent) or other systemic immunosuppressive drugs (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor drugs) within 2 weeks prior to the first medication are allowed to use local, ocular, intra-articular, intranasal, and inhaled corticosteroids
* Subjects with a known history of autoimmune diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, Guillain Barre syndrome, multiple sclerosis, or glomerulonephritis, excluding autoimmune hypothyroidism treated with stable dose hormone replacement therapy
* Individuals with a history of previous immunodeficiency, including those with other acquired or congenital immunodeficiency diseases, or those with a history of organ transplantation, allogeneic bone marrow transplantation, or autologous hematopoietic stem cell transplantation The researcher determined that there are other situations that are not suitable for participation in this study
* The researcher determined that there are other situations that are not suitable for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Cycle 1 of each cohort. Duration of one cycle is 28 days
  DLT is defined as a toxicity (adverse event at least possibly related to LM302) occurring during the DLT observation period
Progression Free Survival (PFS) | From enrollment until 6 months after the last participant discontinues treatment, up to approximately 42 months
  PFS was defined as the time from date of randomization until first objective radiographic tumor progression or death from any cause, based on Investigator assessment

SECONDARY OUTCOMES:
Overall Survival (OS) | From enrollment until 6 months after the last participant discontinues treatment, up to approximately 42 months.
  OS was defined defined as the time from date of randomization until death from any cause.
Objective response rate (ORR) | From start of treatment to date of documented disease progression, up to approximately 42 months
  defined as the proportion of participants who achieve a best response of complete response (CR) or partial response (PR) using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria as assessed by Investigator.
Duration of response (DoR) | From start of treatment to date of documented disease progression, up to approximately 42 months
  defined time from the initial response (CR or PR) until documented tumor progression or death from any cause and based on Investigator assessment.
Disease control rate (DCR) | From start of treatment to date of documented disease progression, up to approximately 42 months
  defined as the proportion of participants who achieved CR, PR, or stable disease (SD) for a minimum of 6 weeks during study treatment, based on Investigator assessment.
. AE and SAE | : From signing the ICF until 28 days after EOT or accept other anti-cancer therapy,up to 40 days after last study dose
  Adverse events will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Tianshu Liu, Doctor, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China